CLINICAL TRIAL: NCT04700800
Title: Regulation of Muscle Protein Phenotype in Humans With Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Lori R. Roust, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 20-003294; R01DK123441 (NIH)
Record Dates: First submitted 2020-12-21; First posted 2021-01-08 (Actual); Results first posted 2025-11-05 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-09

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Subjects with obesity (Experimental): Exercise followed by infusion of amino acids
  Interventions: Other: Exercise
- Lean Subjects (Active Comparator): Exercise followed by infusion of amino acids
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Exercise at 65% of heart rate reserve

SUMMARY:
A hallmark of muscle changes in obesity is an altered muscle fiber type profile, characterized by a reduced proportion of Type I fibers - a shift associated with adverse obesity-related health outcomes. This alteration can be linked to changes in the expression of myosin heavy chain (MHC) protein isoforms in the skeletal muscle of individuals with obesity. The investigators aim to modulate the metabolism of muscle MHC isoforms to uncover the biological mechanisms underlying this disrupted expression pattern in muscle of humans with obesity.

DETAILED DESCRIPTION:
Humans with obesity have typically lower proportion of Type I muscle fibers in skeletal muscle. These fiber types, known for their high capacity for glucose uptake, have also greater sensitivity to fuel metabolism compared with Type II fibers, even within the adverse metabolic environment of obesity. Altered expression of skeletal muscle myosin heavy chain (MHC) protein isoforms, molecular marker of fiber types, may explain this shift.

This project aims to uncover the biological mechanisms sustaining disrupted MHC protein metabolism in the skeletal muscle of individuals with obesity. The investigators will compare overall protein metabolism between humans with obesity and lean controls, with a specific focus on MHC isoforms. They will assess MHC isoform gene expression, associated molecular regulators, and synthesis rates of the MHC isoforms involved in muscle fiber programming. Acute aerobic exercise and elevated plasma amino acids will be used as experimental tools to target transcriptional and translational processes related to MHC gene expression. The findings are expected to reveal mechanisms responsible for the unfavorable fiber type profile observed in the skeletal muscle of humans with obesity.

ELIGIBILITY:
Inclusion Criteria:

* ability to sign informed consent form
* body mass index (BMI), 18-26 kg/m2 (lean subjects), 32-50 kg/m2 (subjects with obesity)

Exclusion Criteria:

* prescription or over-the-counter medication
* supplements known to affect protein metabolism (i.e., amino acids, protein, omega-3 fatty acids)
* diabetes
* acute illness
* liver disease
* uncontrolled metabolic disease, including renal disease
* heart disease related to atrial fibrillation, history of syncope, limiting or unstable angina, congestive heart failure or ECG documented abnormalities
* low hemoglobin or hematocrit
* use of anabolic steroids or corticosteroids (within 3 months)
* not classified as inactive/sedentary based on the Stanford Brief Activity Survey and accelerometry data
* participation in a weight-loss regimen
* extreme dietary practices (i.e., vegan, vegetarian)
* smoking
* pregnancy
* gastro-intestinal surgery
* any other condition or event considered exclusionary by the PI and the study physician.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2021-10-07 (Actual); Primary Completion 2024-10-02 (Actual); Study Completion 2024-10-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lori R Roust, MD, Principal Investigator — Mayo Clinic; Christos S Katsanos, PhD, Principal Investigator — Arizona State University
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 48 participants signed informed consent.
Pre-assignment Details: Of the participants that signed the consent form, 10 were screen failures, 11 withdrew, 4 declined participation, and 1 was enrolled but did not proceed. Twenty-three completed the entire study with one participant had data collected as did part of the study, for a total of 22 with data collected.
Groups:
- Participants with Obesity: Participants with Obesity performing acute aerobic exercise followed by infusion of amino acids, with measurements take before and after exercise+amino acid infusion
- Lean participants: Healthy lean participants performing acute aerobic exercise followed by infusion of amino acids, with measurements take before and after exercise+amino acid infusion
Period: Overall Study
Arm/Group | Participants with Obesity | Lean participants
Started | 10 | 12
Completed | 10 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Lean paticipants: Healthy lean participants performing acute aerobic exercise followed by infusion of amino acids, with measurements take before and after exercise+amino acid infusion
- Total: Total of all reporting groups
Arm/Group | Participants with Obesity | Lean paticipants | Total
Number analyzed (Participants) | 10 | 12 | 22
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age
  Years | 30 (2) | 29 (2) | 29 (2)
Sex: Female, Male [Count of Participants; unit: Participants] — Sex
  Participants
    Female | 6 | 7 | 13
    Male | 4 | 5 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Hispanic/Non-Hispanic
  Participants
    Hispanic or Latino | 1 | 3 | 4
    Not Hispanic or Latino | 9 | 9 | 18
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 8 | 11 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Whole-Muscle Protein Synthesis
Description: Protein synthesis rates in whole muscle were quantified as the fractional synthesis rate (FSR), expressed as %/hour - representing the percentage of the entire muscle protein pool newly synthesized per hour.
  Protein synthesis rates were determined by continuous infusion of a stable isotope-labeled amino acid tracer, followed by measurement of tracer incorporation into the muscle proteins over time.
  Changes in FSR from baseline were evaluated in response to combined exercise and amino acid infusion.
Time Frame: 9 Hours
Measure: Mean (Standard Deviation); unit: %/hr
Arm/Group | Participants with Obesity | Lean participants
Number analyzed (Participants) | 10 | 12
%/hr | 0.004 (0.011) | 0.015 (0.005)

2. Primary Outcome: Synthesis Rates of the Three Myosin Heavy Chain Isoforms (MHC I, MHC IIa, and MHC IIx)
Description: Synthesis rates of the myosin heavy chain protein isoforms were quantified as the fractional synthesis rate (FSR), expressed as %/hour - representing the percentage of each of the three myosin heavy chain isoform protein pool newly synthesized per hour.
  Protein synthesis rates were determined by continuous infusion of a stable isotope-labeled amino acid tracer, followed by measurement of tracer incorporation into each of the three myosin heavy chain isoform protein
  Changes in FSR from baseline were evaluated in response to combined exercise and amino acid infusion.
Time Frame: 9 Hours
Measure: Mean (Standard Deviation); unit: %/hr
Arm/Group | Participants with Obesity | Lean participants
Number analyzed (Participants) | 10 | 12
%/hr
  Myosin Heavy Chain - I (MHC-I) | 0.005 (0.001) | 0.006 (0.001)
  Myosin Heavy Chain -IIa (MHC-IIa) | 0.004 (0.001) | 0.005 (0.001)

3. Primary Outcome: Messenger RNA (mRNA) Expression of Three Myosin Heavy Chain Isoforms (MHC I, MHC IIa, and MHC IIx)
Description: Messenger RNA (mRNA) expressions of the myosin heavy chain isoforms were determined by measuring the abundance of the three specific transcripts of the myosin heavy chain isoforms.
  mRNA was measured using quantitative reverse transcription PCR (qRT-PCR).
  Changes in mRNA expression from baseline were evaluated in response to combined exercise and amino acid infusion.
Time Frame: 9 Hours
Measure: Mean (Standard Deviation); unit: Arbitrary Units
Arm/Group | Participants with Obesity | Lean participants
Number analyzed (Participants) | 10 | 12
Arbitrary Units
  MHC-I | 1.1 (0.5) | 1.0 (0.4)
  MHC-IIa | 0.5 (0.2) | 0.6 (0.3)

ADVERSE EVENTS:
Time Frame: Up to 6 months after enrollment in the study.
Description: Levels of adverse events were defined as: Mild, Moderate, Severe (severe would correspond to serious)
Arm/Group | Participants with Obesity | Lean participants
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/12
Other Adverse Events (participants affected / at risk) | 2/10 | 6/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants with Obesity (N=10) | Lean participants (N=12)
Numbness and soreness on the site of muscle biopsy few days after the procedure (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Nauseous and/or lightheaded (Nervous system disorders) | 0 (0) | 3 (3)
Numbness in mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Unable to drink the drink provided for the oral glucose tolerance test (Gastrointestinal disorders) | 1 (1) | 0 (0)
Car accident outside the study procedures, preventing further participation in the study (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-02-23): https://cdn.clinicaltrials.gov/large-docs/00/NCT04700800/Prot_SAP_001.pdf
  • Informed Consent Form (2024-06-14): https://cdn.clinicaltrials.gov/large-docs/00/NCT04700800/ICF_000.pdf